CLINICAL TRIAL: NCT02305602
Title: A Phase I, Open-label Study of the Effects of Percutaneous Administration of an Extracellular Matrix Hydrogel, VentriGel, Following Myocardial Infarction
Brief Title: A Study of VentriGel in Post-MI Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ventrix, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CV-201
Record Dates: First submitted 2014-11-26; First posted 2014-12-02 (Estimated); Last update posted 2019-10-25 (Actual); Status verified 2019-10

CONDITIONS: Myocardial Infarction; Heart Failure; Left Ventricular Remodeling
Keywords: extracellular matrix
MeSH Terms: conditions — Myocardial Infarction; Heart Failure; Ventricular Remodeling

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Post Myocardial Infarction (Experimental): VentriGel will be injected via a MyoStar catheter after NOGA mapping in the 60 day to 3 year window since the first STEMI myocardial infarction
  Interventions: Biological: VentriGel

INTERVENTIONS:
Biological: VentriGel — VentriGel will be injected via MyoStar catheter after NOGA mapping

SUMMARY:
This Phase I, open label, study will investigate the effects of VentriGel injection in patients who have experienced a first, large ST elevation myocardial infarction (STEMI) treated by PCI within the past 3 years and have evidence of left ventricular remodeling.

DETAILED DESCRIPTION:
Evaluate the safety and feasibility of VentriGel delivered trans-endocardially to subjects with left ventricular ejection fraction (LVEF) 25 to 45% secondary to MI. Secondary endpoints will look at efficacy variables of ESV, EDV, EF, scar mass.

ELIGIBILITY:
Inclusion Criteria:

1. The subject is 30-75 years of age
2. The subject must be able to provide informed consent
3. At least 60 days and no more than 3 years will have passed since the first ST elevation myocardial infarction (Index STEMI) at time of VentriGel administration
4. The Index STEMI must meet the following criteria:

   1. First time diagnosis of STEMI AND;
   2. Meet the STEMI criteria of the American College of Cardiology (ACC)/American Heart Association (AHA) (e.g. ST elevation in at least 2 contiguous leads >0.2 mV in V1, V2 or V3 and/or >0.1mV in at least two other leads), or new left bundle branch block (LBBB)
5. Evidence of left ventricular remodeling secondary to the myocardial infarction using 2-D echocardiography or cMR;

   1. the LVEF must be ≥ 25% and ≤ 45% AND;
   2. The left ventricular wall thickness is ≥ 8 mm in target area.
6. Successful percutaneous coronary intervention (PCI) restoring TIMI II of higher flow to infarcted area
7. Negative pregnancy test [serum human chorionic gonadotropin (βhCG)] in women of childbearing potential within 24 hours prior to dosing) or if less than 2 years postmenopausal agree to use of adequate contraception during the study.
8. Must be ambulatory, willing and able to comply with protocol, including follow-up visits
9. Subject must be receiving best medical treatment for their post-MI clinical presentation according to the American College of Cardiology (ACC)/American Heart Association (AHA) guidelines
10. For those subjects indicated for heart failure medical therapy, subjects must be on stable therapy including beta-blockers and angiotensin converting enzyme inhibitors, if tolerated, for at least 45 days prior to therapy delivery

Exclusion Criteria:

1. Contraindications to cardiac MR
2. NYHA Functional Classification 4 heart failure within the prior 6 months.
3. Significant coronary artery stenosis that may require percutaneous or surgical revascularization within six months of enrollment, as determined by the principal investigator
4. Left ventricular thrombus, left ventricular aneurysm, subjects with post-infarction pericarditis, or subjects with wall motion abnormalities outside the region of the infarct related artery
5. Frequent, recurrent, sustained (>30 seconds) ventricular tachycardia in 30 days prior to VentriGel administration
6. ECG or 24 hour Holter Monitor with any of the following findings:

   * Bifascicular block (left bundle branch block or right bundle branch block plus left hemi-block)
   * Higher grade AV block (i.e. 3rd degree)
   * Ventricular tachycardia (>= 5 seconds of VT OR any symptomatic VT)
7. Atrial fibrillation with heart rate greater than 110 bpm.
8. Severe valvular disease (e.g. aortic stenosis of moderate or worse severity, valvular insufficiency requiring surgical repair) or history of heart valve replacement.
9. Known allergy to porcine proteins or prior implantation of a porcine derived medical product including cardiac valves or other ECM products.
10. Etiology of heart failure due to any cause (e.g. hypertrophic cardiomyopathies, restrictive cardiomyopathies, constrictive pericardial disease, amyloidosis, active myocarditis) other than the index MI.
11. Severe peripheral vascular disease that impairs femoral arterial access.
12. Less than 3 years, cancer free, since end of treatment for cancer (with exception of basal cell carcinoma)
13. Alcohol or drug dependency within six months prior to enrollment
14. Cerebrovascular event within the 90 days prior or major surgical procedure or major trauma within the 14 days prior to enrollment
15. Participation, defined as receiving test article, in an experimental clinical study within 30 days prior to administration of VentriGel (i.e. screen failure from other study does not exclude subject)
16. Uncontrolled hypertension defined as systolic blood pressure (SBP) > 180 mmHg and/or or diastolic blood pressure (DBP) >110 mmHg
17. Abnormal laboratory values as defined below performed at screening:

    * Aspartate aminotransferase [AST]/ alanine aminotransferase [ALT] ≥ 3 times upper limit of normal (ULN)
    * Serum creatinine ≥ 2.0 mg/dL
    * Platelet count < 50,000/mm3
    * Hemoglobin < 9.0 g/dL
    * HbA1c > 9.0%
    * PT or aPTT with clinically significant elevations relative to local laboratory norms
18. Any other cardiac or non-cardiac conditions or illness which, in the opinion of the principal investigator, may place subjects at undue risk or compromise the objectives of the study.
19. Institutional interpretation of cMR EF data outside the ≥ 25% and ≤ 45% limits

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2018-09-05 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Incidence of serious adverse events that occur within 6 months of injection | 6 months

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Mercy Gilbert Medical Center, Gilbert, Arizona
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of Florida, Gainesville, Florida
  - Rush University Medical Center, Chicago, Illinois
  - Minneapolis Heart Institute, Minneapolis, Minnesota
  - University of Utah, Salt Lake City, Utah